CLINICAL TRIAL: NCT04998123
Title: A Randomized, Sham-controlled Study of the Efficacy of Intersectional Short Pulse (ISP) Stimulation for Seizure Termination
Brief Title: Efficacy of Intersectional Short Pulse Stimulation for Terminating Seizures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not receive funding for the study.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-00698
Record Dates: First submitted 2021-08-04; First posted 2021-08-10 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Seizures; Focal Epilepsy
MeSH Terms: conditions — Seizures; Epilepsies, Partial

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The subject will be blinded to the treatment condition. The study team clinician will be aware of the treatment condition to provide to the clinical team any necessary information for clinical care. Decisions by expert review of EEG on seizure duration will be blinded to treatment condition as well.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Sham Stimulation (Sham Comparator)
  Interventions: Device: SeizureStop Device
- ISP Stimulation (Experimental)
  Interventions: Device: SeizureStop Device
- Perpheral Stimulation (No Intervention)

INTERVENTIONS:
Device: SeizureStop Device — Intersectional Short Pulse (ISP) Stimulation will be performed using SeizureStop Device. The ISP stimulation method proposed in this study is to increase the intensity of stimulation delivered to targeted brain regions, while minimizing the peripheral effects of stimulation. For sham stimulation, no settings will be modified.
  Arms: ISP Stimulation; Sham Stimulation

SUMMARY:
This is a study which seeks to develop a novel therapeutic approach, Intersectional Short Pulse (ISP) stimulation for seizure termination. The device embodiment of ISP is a scalp EEG recording system which also delivers spatially precise electrical stimulation in short pulses to the targeted brain region. The study team has already collected safety and tolerability data in human subjects, demonstrated ISP efficacy in terminating seizures in rodents, and have tested the efficacy of this device to modulate normal human brain activity. Now this study proposes to test the device's efficacy in stopping seizures in a within-subject randomized, sham-controlled study design.

ELIGIBILITY:
Experiment 3: Epilepsy patients

Inclusion criteria:

* Adult patients (age 18-65).
* Fluent in English.
* Epilepsy patients with poorly controlled (>=2 seizures per week).
* Focal onset seizures.
* Seizure onset zone in the mesial temporal or neocortical onset as determined by >2 concordant criteria, without discordant criteria (semiology, MRI Brain, and EEG).
* Able to give informed consent.

Exclusion criteria:

* Patients with skull defects.
* Patients with implanted neurostimulator or other implanted cerebral hardware.
* Patients with multifocal onset epilepsy.
* Patients who are non-verbal or incapable of providing informed consent.
* Current substance abuse.
* Pregnancy.
* Patients with non-MRI compatible implants (for Experiments 2 and 3).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Mean duration of seizures detected | up to Day 10

CONTACTS AND LOCATIONS:
Overall Officials: Anli Liu, MD, MA, Principal Investigator — NYU Langone Health

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal will have access to the data upon reasonable request. Data are available for 5 years at a third party website (Link to be included).